CLINICAL TRIAL: NCT05776940
Title: Probiotic Supplementation Reduces Gastrointestinal Symptoms During the Therapy and Improves Therapeutic Response in AL Amyloidosis: A Randomized Controlled Trial
Brief Title: Probiotic Supplementation Reduces Gastrointestinal Symptoms During the Therapy and Improves Therapeutic Response in AL Amyloidosis
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Shiren sun, Professor, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Probiotic in AL amyloidosis
Record Dates: First submitted 2023-02-08; First posted 2023-03-20 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Immunoglobulin Light-chain Amyloidosis
MeSH Terms: conditions — Immunoglobulin Light-chain Amyloidosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic group (Active Comparator): Naive al amyloidosis patients receive Bortezomib+Dexamethasone, Bortezomib+Dexamethasone+Daratumumab or single Daratumumab therapy combined with Live Combined Bacillus Subtilis and Enterococcus Faecium Enteric-coated Capsules( 250mg/time, bid,up to 3 months).
  Interventions: Drug: Live Combined Bacillus Subtilis and Enterococcus Faecium Enteric-coated Capsules combined with Bortezomib+Dexamethasone/Bortezomib+Dexamethasone+Daratumumab/single Daratumumab
- Control group (Active Comparator): Naive al amyloidosis patients receive Bortezomib+Dexamethasone, Bortezomib+Dexamethasone+Daratumumab or single Daratumumab therapy without any probiotics.
  Interventions: Drug: Bortezomib+Dexamethasone/Bortezomib+Dexamethasone+Daratumumab/single Daratumumab

INTERVENTIONS:
Drug: Live Combined Bacillus Subtilis and Enterococcus Faecium Enteric-coated Capsules combined with Bortezomib+Dexamethasone/Bortezomib+Dexamethasone+Daratumumab/single Daratumumab — Naive al amyloidosis patients receive Bortezomib+Dexamethasone, Bortezomib+Dexamethasone+Daratumumab or single Daratumumab therapy combined with Live Combined Bacillus Subtilis and Enterococcus Faecium Enteric-coated Capsules(250mg/time, bid,up to 3 months).
  Other Names: Live Combined Bacillus Subtilis and Enterococcus Faecium Enteric-coated Capsules + Routine therapy
  Arms: Probiotic group
Drug: Bortezomib+Dexamethasone/Bortezomib+Dexamethasone+Daratumumab/single Daratumumab — Naive al amyloidosis patients receive Bortezomib+Dexamethasone, Bortezomib+Dexamethasone+Daratumumab or single Daratumumab therapy without any probiotics (Blank Control).
  Other Names: Routine therapy
  Arms: Control group

SUMMARY:
The purpose of this clinical trial is to evaluate whether specific probiotic can reduce gastrointestinal symptoms and improves therapeutic response, on a background of Bortezomib+dexamethasone or Bortezomib+dexamethasone combined with daratumumab therapy, for naive AL amyloidosis patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Biopsy-proven naive AL amyloidosis
* Receive at least 1 course of treatment based on Bortezomib+Dexamethasone or Bortezomib+Dexamethasone+Daratumumab therapy
* At least 1 organ (heart, kidney, liver, etc) involved
* Agree to participate in the project and sign the informed consent.

Exclusion Criteria:

* Received antibiotics for 3 consecutive days and on in the past 2 months prior to the enrollment
* Had history of probiotics, prebiotics, immunosuppressants, hormones, and other medications use in the past 3 months that influence the Gastrointestinal Microbiome
* Had other underlying diseases（malignancy or immune system diseases, etc.）
* Had history of clearly diagnosed chronic gastrointestinal disease
* Secondary AL amyloidosis or local AL amyloidosis
* Other conditions the researcher judged unsuitable for enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2023-03-31 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Occurrence of diarrhea | Up to 3 months after enrollment
  Increased stool frequency and/or loose or watery stools

SECONDARY OUTCOMES:
Time before diarrhea | Up to 3 months after enrollment
  Time interval from the start of treatment to the first diarrhea
Duration of the diarrhea | Up to 6 months after enrollment
  The time between the start of diarrhea and the last diarrhea.
Hematological response at 3 and 6 months after enrollment | Up to 6 months after enrollment
  Hematological response is evaluated according to the difference between Serum free light chains and immunofixation electrophoresis.
Involved organ response（heart）at 3 and 6 months after enrollment | Up to 6 months after enrollment
  Involved organ response（heart）is evaluated according to the change of NT-proBNP.
SF-36 score at 1 month, 3 month and 6 month | Up to 6 months after enrollment
  The general health condition is evaluated by the 36-item Short-Form. The SF-36 measure consists of 36 items that address the following 8 dimensions: physical pain, mental health, general health, emotional role functioning, social functioning, vitality, and physical and role functioning. Each dimension receives a final score between 0 and 100, with 100 representing the best performance.
GSRS score at 1 month, 3 month and 6 month | Up to 6 months after enrollment
  The Gastrointestinal Symptoms are evaluated by Gastrointestinal Symptom Rating Scale. The minimum and maximum values is 15 and 105, respectively. The scores are calculated by taking the mean of the items completed within an individual scale, with higher scores indicating greater severity of symptoms.
Other adverse events that occurred during the treatment | Up to 6 months after enrollment
  Adverse events are evaluated according to the CTCAE 5.0.
Survival status at study endpoints | From date of randomization until the date of death from any cause, assessed up to 36 months
  Survival status（live or dead）
Changes of al amyloidosis patients' gut microbiome at 3 months and 6 months after enrollment | Up to 6 months after enrollment.
  The changes of gut microbiome are evaluated by 16sRNA (such as Microbiota α-diversity and β-diversity、Changes in gut microbiota at the phylum and the genus levels、Phylogenetic profiles of the gut microbial communities、Microbial functional alteration、Correlations between significantly different ASVs and clinical characteristics in AL amyloidosis patients.etc.)
Severity of the diarrhea | Up to 6 months after enrollment
  The severity of diarrhea was graded according to the CTCAE 5.0.
Involved organ response（kidney）at 3 and 6 months after enrollment | Up to 6 months after enrollment
  Involved organ response（kidney）is evaluated according to the change of 24h proteinuria.